CLINICAL TRIAL: NCT04863456
Title: Efficiency and Safety of Different Treatment Strategies in Adults With Pituitary Adenomas With Hypothalamic Involvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2021]IEC-J(227)
Record Dates: First submitted 2021-03-29; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Pituitary Adenoma
Keywords: pituitary adenoma; treatment strategy; Hypothalamus
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIPA group of Puget grade 1 (Experimental): the tumor abuting or displacing the hypothalamus in the preoperative MR images
  Interventions: Procedure: Total resection; Procedure: Staged resection; Procedure: Subtotal resection followed by stereotactic radiation therapy
- HIPA group of Puget grade 2 (Experimental): hypothalamic involvement (the hypothalamus is no longer identifiable) in the preoperative MR images
  Interventions: Procedure: Total resection; Procedure: Staged resection; Procedure: Subtotal resection followed by stereotactic radiation therapy

INTERVENTIONS:
Procedure: Total resection — Total resection of HIPA in a single surgery
Procedure: Staged resection — HIPA was resected subtotally at first time, and the tumor remnant was removed at a later date
Procedure: Subtotal resection followed by stereotactic radiation therapy — HIPA was resected subtotally at first time, and the tumor remnant was controled by the stereotactic radiation therapy

SUMMARY:
Prospective and randomized evaluate efficiency and safety of different treatment strategies for hypothalamus-invading pituitary adenomas (HIPA)

DETAILED DESCRIPTION:
There are various treatment strategies for hypothalamus-invading pituitary adenomas (HIPA), such as total resection (TR), subtotal resection with radiosurgery (STR+RS), etc. However,the optimal treatment of HIPA is still controversial. In this study, we want to evaluate the efficiency and safety of different treatment strategies in adults with HIPA.

ELIGIBILITY:
Inclusion Criteria:

* Suspected symptomatic or progressively growing pituitary adenoma with Hypothalamic Involvement
* Informed consent

Exclusion Criteria:

* No follow-up possible
* Emergency surgery without informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of QoL (Quality of Life, EQ-5D) for the first surgery | baseline (before the first surgery), 2 years after the first surgery
  EQ-5D will be evaluated before the first surgery and after the first surgery in 2 years
Change of QoL (Quality of Life, EQ-5D) for the second intervention | baseline (before the second intervention), 3 months after the second intervention
  EQ-5D will be evaluated before the second intervention and after the second intervention in 3 months

SECONDARY OUTCOMES:
Change of Visual Acuity statue | baseline (before the first surgery), 2 years after the first surgery
  Visual Acuity statue will be evaluated using Snellen's chart before the first surgery and after the first surgery in 2 years
Change of Visual Field statue | baseline (before the first surgery), 2 years after the first surgery
  Visual Field statue will be evaluated using a Humphrey visual field analyser before the first surgery and after the first surgery in 2 years
Change of Hormone Replacement Therapy | baseline (before the first surgery), 2 years after the first surgery
  Whether the Hormone Replacement Therapy was used (Yes or No) before the first surgery and after the first surgery in 2 years
Extent of resection | baseline (before the first surgery), 2 years after the first surgery
  Volumetric analysis of tumor volume before the first surgery, intraoperatively and 3 months and 2 years after the first surgery will be performed. In addition, Tumor volume will be evaluated before the second intervention and intraoperatively. Gross total resection is defined as no tumor present in gadolinium enhanced T1 sequences.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Huang, PhD, MD, Study Director — Department of Neurosurgery, Union hospital, Huazhong University of Science and Technology